CLINICAL TRIAL: NCT01923220
Title: An Open-Label, Randomized Study to Evaluate the Safety and Efficacy of HO/02/02 20µg vs. SoC (Aloe Vera) to Reduce Radiation Dermatitis In Breast Cancer Patients Undergoing Radiation Therapy.
Brief Title: Safety and Efficacy of HO/02/02 20µg vs. SoC (Aloe Vera) to Reduce Radiation Dermatitis
Acronym: ARD
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HealOr (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HO-ARD-01-2012
Record Dates: First submitted 2013-08-12; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Radiation Therapy; Radiation Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HO/02/02 (Experimental): Interventions involving HO/02/02 20µg VS. Aloe Vera Jel (SOC). Treatment will be applied topically once daily
  Interventions: Drug: HO/02/02 20µg
- Aloe Vera Jel (Sham Comparator): To be applied topically
  Interventions: Other: Aloe Vera Jel

INTERVENTIONS:
Drug: HO/02/02 20µg — Interventions involving HO/02/02 20µg VS. Aloe Vera Jel (SOC). Treatment will be applied topically once daily
  Arms: HO/02/02
Other: Aloe Vera Jel — To be applied topically once daily
  Arms: Aloe Vera Jel

SUMMARY:
This is a single-center, open-label, randomized, prospective study evaluating the safety and efficacy of HO/02/02 20µg topically applied daily for 15 minutes (with gauze) on treatment fields vs. standard of care (SoC), Aloe Vera treatment

DETAILED DESCRIPTION:
This is a single-center, open-label, randomized, prospective study evaluating the safety and efficacy of HO/02/02 20µg topically applied daily for 15 minutes (with gauze) on treatment fields vs. standard of care (SoC), Aloe Vera treatment in addition to sterile water for irrigation applied daily for 15 minutes (with gauze) on treatment fields to create the same cooling effect as in treatment arm 1. Both treatment arms 1&2 treatments will be applied topically once daily for up to 8 weeks to reduce radiation dermatitis in up to 90 breast cancer patients undergoing adjuvant radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years old and above.
* Histology confirmed unilateral breast cancer following lumpectomy
* Planned to receive 50 Gy, whole breast XRT and regional lymph nodes radiation.
* ECOG performance status 0-2
* Completed Chemotherapy 3 weeks prior to XRT (if applicable)
* Patient should be available for the entire study period, and be able and willing to adhere to protocol requirements;
* Patient must sign an informed consent form prior to undergoing any study-related procedures

Exclusion Criteria:

* Known uncontrolled diabetes
* Prior radiation to breast
* Known connective tissue disorder
* Known skin disease over the treated breast
* Prior burn over treated area
* Evidence of infection or inflammation of breast to be treated.
* Receiving biological therapy or hormone therapy (other than Herceptin) during radiation treatment/study duration and 4 weeks prior to study entry.
* Pre-existing skin breakdown within the planned radiotherapy field at the time of study entry.
* Pregnancy, planned pregnancy, lactation or inadequate contraception as judged by the Investigator.
* Participation in another investigational drug or vaccine trial concurrently or within 30 days.
* Use of any other topical or systemic treatments aimed at radiation dermatitis.
* Use of a prescription or over-the-counter medication that contains hydrocortisone or any other cortisone or corticosteroid containing preparation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients using HO/02/02 20µg that developed grade 1-4 radiation dermatitis during adjuvant radiation therapy for breast cancer compared to SoC (Aloe Vera) commonly used as standard of care treatment. | 62 days

SECONDARY OUTCOMES:
Frequency and severity of adverse events reported by the patients and assessed clinically by NCI CTC v2.0 | 62 Days

CONTACTS AND LOCATIONS:
Overall Officials: Yair Alegranti, Study Director — HealOr
Locations (1):
- The Chaim Sheba Medical Center, Ramat Gan, Israel